CLINICAL TRIAL: NCT06563908
Title: Lipiodol® For Enhancing Live Birth Rates In Infertile Couples Undergoing In Vitro Fertilization/ Intracytoplasmic Sperm Injection A Randomized Controlled Trial
Brief Title: Lipiodol Prior to FET (LIFE)
Acronym: LIFE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1767/QD-BYT
Record Dates: First submitted 2024-08-01; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: IVF; Frozen Embryo Transfer; Hysterosalpingography
Keywords: Lipiodol; Hysterosalpingography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipiodol® uterine treatment prior to IVF/ICSI (Experimental): For those who are randomized to Lipiodol®, treatment will be performed by a HSG technique with X-ray screening on day 3 or day 5 after oocyte retrieval. The contrast medium will be Lipiodol Ultra Fluide® (Guerbet, France), an iodized poppy seed oil obtained by substitution of ethyl esters for the glyceryl esters of Lipiodol®. After that the procedure to assess study participants' pain perception.
  Endometrial preparation for frozen embryo transfer will perform on the subsequence cycle
  Interventions: Procedure: Lipiodol® uterine treatment prior to IVF/ICSI
- No Lipiodol® uterine treatment prior to IVF/ICSI (No Intervention): For those who are randomized to no intervention arm (control group), there will be no HSG performed.
  Endometrial preparation for frozen embryo transfer will perform on the subsequence cycle

INTERVENTIONS:
Procedure: Lipiodol® uterine treatment prior to IVF/ICSI — Lipiodol®, treatment will be performed by a HSG technique with X-ray screening on day 3 or day 5 after oocyte retrieval. The contrast medium will be Lipiodol Ultra Fluide® (Guerbet, France), an iodized poppy seed oil obtained by substitution of ethyl esters for the glyceryl esters of Lipiodol®. One millilitre of Lipiodol Ultra Fluide® contains 0.48g iodine. Women will lie in the left lateral or supine position. Radiologists will use a 'no touch' technique after applying antiseptic solution to the cervix. Uterine cannulation using the Cook HSG catheter will be applied to conduct Lipiodol® treatment. Prewarmed (37oC) Lipiodol® will be slowly instilled, with intermittent fluoroscopic X-ray guidance. Up to 10 ml of Lipiodol® will be slowly injected into the uterus and directly monitored by fluoroscopy. If intravasation was observed on X-ray (contrast apparent in the venous system), instillation will be stopped immediately.
  Other Names: Lipiodol® flushing prior to IVF/ICSI
  Arms: Lipiodol® uterine treatment prior to IVF/ICSI

SUMMARY:
Lipiodol® flushing is an effective fertility treatment for women with unexplained infertility. It is speculated that the treatment effect could work through a direct effect of Lipiodol® on the endometrium. Given this direct effect on the endometrium, it is further hypothesized that Lipiodol® uterine treatment prior to In Vitro Fertilization (IVF)/ Intracytoplasmic Sperm Injection (ICSI) may also improve pregnancy rates. However, the effectiveness of Lipiodol® as an adjunct to IVF/ICSI treatment has not previously been examined in a well-powered and properly conducted randomised clinical trial.

DETAILED DESCRIPTION:
Study procedures:

Recruitment:

Potentially eligible patients will be given information about the study and a copy of the informed consent documents on day 2 - 3 of their menstrual cycle, when the ovarian stimulation starts. On the day of freeze-all (3 days or 5 days after oocyte retrieval), screening for eligibility will be performed by treating physicians. Eligible couples will have about an hour to decide if they will participate in the study or not. If they choose to participate in the study, investigators will ask them to sign the consent form.

Once a participant signs an informed consent she is enrolled in the study. An individual record of all non-recruited patients and reasons for exclusion (at any stage) will be obtained and stored

Randomization:

Assignment to treatment allocation will be done via a web portal hosted by Hope Research Center, Viet Nam. The randomisation schedule will be computer-generated at Hope Research Center by using HRC (Hope Research Center) Epi software, in a 1:1 ratio, with a permuted random block size of 4 or 6.

Other standard assisted reproductive treatments are similar and parallel between the two groups, except for the use of Lipiodol® flushing in the intervention group. Due to the type of interventions, this study will only be blinded to clinicians who performed the embryo transfer and embryologists in the IVF clinics.

In the subsequent cycle, all patients in both groups will undergo frozen embryo transfer by using exogenous steroids regimen, starting from day 2 to day 4 of the menstrual cycle. Oral estradiol valerate (Progynova, Bayer Schering Pharma, Germany) 8 mg/day is given for 10-12 days. Ultrasound monitoring will be performed from day tenth onward. When endometrial thickness reaches greater than or equal to 8 mm, along with a triple-line pattern, micronized progesterone 800 mg will be administrated. Frozen embryo transfer (FET) will be performed 3-5 days after progesterone administration, depending on embryo staging. After FET, estradiol and progesterone supplementation are continued for all patients until the day of the pregnancy test. Patients with a positive pregnancy test will continue to receive luteal phase support regimen until 7 weeks of gestation.

All participants will be followed up per local protocol until outcomes are achieved

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF/ICSI
* Having indications for freeze-all (day-3 or day-5)
* Agree to have ≤ 2 frozen embryos transferred
* TSH < 2.5 mIU/mL
* Permanent resident in Viet Nam
* Agree to participate in the study by signing the inform consent

Exclusion Criteria:

* Iodine allergy
* History of salpingectomy or tubal ligation
* History of using Lipiodol® within 6 months prior, starting from the screening time
* At high risk of having Fallopian tube disorders (history of Chlamydia infection, history of pelvic inflammatory diseases, current endometriosis)
* Having evidence of Fallopian tube disorders on Hysterosalpingo - Foam Sonography (HyFoSy), hysterosalpingography (HSG), ultrasonography or laparoscopy
* Having untreated intrauterine lesions such as endometrial polyps, submucosal fibroids, etc which affect the outcome of IVF treatment
* Have a history of thyroid disease or being treated for thyroid disease
* Undergoing curettage within 30 days before performing HSG technique
* Patients having embryos from oocyte donation or in vitro maturation (IVM) cycles
* Unable or unwilling to attend Lipiodol® procedure
* Participating in another interventional study at the same time

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 784 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Live birth rate after the first transfer | At 22 weeks of gestation
  Live birth is defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age, which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. If gestational age is unknown, a birth weight of 500 grams or more will be used instead

SECONDARY OUTCOMES:
Positive pregnancy test | At 2 weeks after embryo(s) placement
  Serum human chorionic gonadotropin level greater than 25 mIU/mL (milli-International Unit per milliliter)
Clinical pregnancy rate | At 5 weeks after embryo(s) placement
  Clinical pregnancy is diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy at 6 weeks or more after the onset of last menstrual period. In addition to intra-uterine pregnancy, it includes a clinically documented ectopic pregnancy
Ongoing pregnancy rate | At 10 weeks after embryo(s) placement
  Ongoing pregnancy is a pregnancy with a detectable heart rate at 12 weeks gestation or beyond
Multiple pregnancy | At 7 weeks after embryo(s) placement
  The presence of more than one gestational sac at early pregnancy ultrasound (6-9 weeks gestation)
Cumulative live birth rate at 12 months after randomization | At 12 months after randomization
  Cumulative live birth at 12 months after randomization
Ectopic pregnancy rate | At 12 weeks of gestation
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology
Early miscarriage rate (Miscarriage <12 weeks) | At 12 weeks of gestation
  A spontaneous loss of pregnancy up to 12 weeks of gestation.
Late miscarriage rate (Miscarriage <22 weeks) | At 22 weeks of gestation
  A spontaneous loss of pregnancy between 12 to 22 weeks.
Still birth rate | After 22 weeks of gestation
  The death of a fetus prior to the complete expulsion or extraction from its mother after 20 completed weeks of gestational age. The death is determined by the fact that, after such separation, the fetus does not breathe or show any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles. It includes deaths occurring during labor
Adverse events | At delivery
  Include intravasation of Lipiodol® and lipogranuloma formation, as well as all other adverse events
Maternal thyroid function | At the day of pregnancy test, 3 months (at 7 weeks of pregnancy if the patient is pregnant) and 6 months (at 22 weeks of pregnancy if the patient is pregnant) after randomization
  Serum TSH and FT4
Gestational diabetes mellitus rate | At 24-28 weeks of gestation
  Using a 75g oral glucose tolerance test, with plasma glucose measurement when patient is fasting and at 1 and 2 h, at 24-28 weeks of gestation in women not previously diagnosed with diabetes.
  * Fasting: 92 mg/dL (5.1 mmol/L)
  * 1 h: 180 mg/dL (10.0 mmol/L)
  * 2 h: 153 mg/dL (8.5 mmol/L)
Hypertensive disorders of pregnancy rate | From date of randomization until the date of first documented progression, assessed up to 12 months after randomization
  Percentage of pregnancy-induced hypertension (PIH), pre-eclampsia (PET), eclampsia, and HELLP syndrome
Preterm birth rate | At 22, 28, 32 and 37 weeks of gestation
  Defined as any delivery at <24, <28, <32, <37 completed weeks' gestation
Premature rupture of membranes rate | At 37 weeks of gestation
  A rupture of the membranes (amniotic sac) prior to 37 weeks' gestation.
Chorioamnionitis rate | At delivery
  Chorioamnionitis is defined as intraamniotic infection with resultant inflammation of any combination of the amniotic fluid, placenta, fetus, fetal membranes, or decidua
Percentage of magnesium sulfate administration for neuroprotection | At delivery
  Administration of magnesium sulfate for preventing seizures in case of preeclampsia/eclampsia
Antenatal corticosteroids for lung maturation | At delivery
  Administration of corticosteroids prior to preterm birth
Administration of tocolytics agents | At delivery
  Administration of tocolytics agents to prevent preterm birth
Birth weight | At delivery
  including low birth weight (defined as weight < 2,500 gram at birth), very low birth weight (defined as < 1,500 gram at birth), high birth weight (defined as >4,000 gram at birth) and very high birth weight (defined as >4,500 gram at birth)
Large for gestational age | At delivery
  Birth weight >90th centile for gestation, based on standardized ethnicity-based charts
Small for gestational age | At delivery
  Birth weight <10th centile for gestation age based on standardized ethnicity-based charts
Gestational age at birth | At delivery
  Calculated by gestational age of all live births
Mode of delivery | At delivery
  including vaginal delivery, C-section (elective, suspected fetal distress, non-progressive labor)
Postpartum hemorrhage | At delivery
  Cumulative blood loss greater than or equal to 1,000 mL or blood loss accompanied by signs or symptoms of hypovolemia within 24 hours after the birth process (includes intrapartum loss) regardless of route of delivery
Maternal death | At delivery
  Female deaths from any cause related to or aggravated by pregnancy or its management (excluding accidental or incidental causes) during pregnancy and childbirth or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy
Congenital anomalies | Within 28 days of birth
  Structural or functional disorders that occur during intra-uterine life and can be identified prenatally, at birth or later in life
Neonatal mortality | Within 28 days of birth
  Death of a live born baby within 28 days of birth
neonatal intensive care unit (NICU) admission | Within 28 days of birth
  The admittance of the newborn to NICU
1-minute Apgar score | At 1 minute after birth
  The Apgar score at 1 minute after birth
5-minute Apgar score | At 5 minute after birth
  The Apgar score at 5 minute after birth
Low 5-minute Apgar score | At 5 minute after birth
  Defined as 5-minute Apgar score <7.
Neonatal thyroid function | At delivery
  Serum thyroid-stimulating hormone (TSH) and free thyroxine (fT4)
Mode of conception | From date of randomization until the date of pregnancy test or date of ultrasound, whichever came first, assessed up to 12 months
  Including natural conception, intrauterine insemination (IUI), and in vitro fertilization (IVF)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thoma ME, McLain AC, Louis JF, King RB, Trumble AC, Sundaram R, Buck Louis GM. Prevalence of infertility in the United States as estimated by the current duration approach and a traditional constructed approach. Fertil Steril. 2013 Apr;99(5):1324-1331.e1. doi: 10.1016/j.fertnstert.2012.11.037. Epub 2013 Jan 3. PMID 23290741
- [Background] Abrao MS, Muzii L, Marana R. Anatomical causes of female infertility and their management. Int J Gynaecol Obstet. 2013 Dec;123 Suppl 2:S18-24. doi: 10.1016/j.ijgo.2013.09.008. Epub 2013 Sep 11. PMID 24119894
- [Background] WEIR WC, WEIR DR. Therapeutic value of salpingograms in infertility. Fertil Steril. 1951 Nov-Dec;2(6):514-22. doi: 10.1016/s0015-0282(16)30725-7. No abstract available. PMID 14887769
- [Background] KING EL, HERRING JS. Sterility studies in private practice. Am J Obstet Gynecol. 1949 Aug;58(2):258-66. doi: 10.1016/0002-9378(49)90378-6. No abstract available. PMID 18133559
- [Background] Watson A, Vandekerckhove P, Lilford R, Vail A, Brosens I, Hughes E. A meta-analysis of the therapeutic role of oil soluble contrast media at hysterosalpingography: a surprising result? Fertil Steril. 1994 Mar;61(3):470-7. doi: 10.1016/s0015-0282(16)56578-9. PMID 8137969
- [Background] Mohiyiddeen L, Hardiman A, Fitzgerald C, Hughes E, Mol BW, Johnson N, Watson A. Tubal flushing for subfertility. Cochrane Database Syst Rev. 2015 May 1;2015(5):CD003718. doi: 10.1002/14651858.CD003718.pub4. PMID 25929235
- [Background] Dreyer K, van Rijswijk J, Mijatovic V, Goddijn M, Verhoeve HR, van Rooij IAJ, Hoek A, Bourdrez P, Nap AW, Rijnsaardt-Lukassen HGM, Timmerman CCM, Kaplan M, Hooker AB, Gijsen AP, van Golde R, van Heteren CF, Sluijmer AV, de Bruin JP, Smeenk JMJ, de Boer JAM, Scheenjes E, Duijn AEJ, Mozes A, Pelinck MJ, Traas MAF, van Hooff MHA, van Unnik GA, de Koning CH, van Geloven N, Twisk JWR, Hompes PGA, Mol BWJ. Oil-Based or Water-Based Contrast for Hysterosalpingography in Infertile Women. N Engl J Med. 2017 May 25;376(21):2043-2052. doi: 10.1056/NEJMoa1612337. Epub 2017 May 18. PMID 28520519
- [Background] Johnson JV, Montoya IA, Olive DL. Ethiodol oil contrast medium inhibits macrophage phagocytosis and adherence by altering membrane electronegativity and microviscosity. Fertil Steril. 1992 Sep;58(3):511-7. doi: 10.1016/s0015-0282(16)55254-6. PMID 1325928
- [Background] Sawatari Y, Horii T, Hoshiai H. Oily contrast medium as a therapeutic agent for infertility because of mild endometriosis. Fertil Steril. 1993 Apr;59(4):907-11. doi: 10.1016/s0015-0282(16)55880-4. PMID 8384577
- [Background] Mikulska D, Kurzawa R, Rozewicka L. Morphology of in vitro sperm phagocytosis by rat peritoneal macrophages under influence of oily contrast medium (Lipiodol). Acta Eur Fertil. 1994 May-Jun;25(3):203-6. PMID 7900503
- [Background] Johnson NP, Farquhar CM, Hadden WE, Suckling J, Yu Y, Sadler L. The FLUSH trial--flushing with lipiodol for unexplained (and endometriosis-related) subfertility by hysterosalpingography: a randomized trial. Hum Reprod. 2004 Sep;19(9):2043-51. doi: 10.1093/humrep/deh418. Epub 2004 Jul 22. PMID 15271870
- [Background] Johnson NP, Bhattu S, Wagner A, Blake DA, Chamley LW. Lipiodol alters murine uterine dendritic cell populations: a potential mechanism for the fertility-enhancing effect of lipiodol. Fertil Steril. 2005 Jun;83(6):1814-21. doi: 10.1016/j.fertnstert.2004.11.065. PMID 15950655
- [Background] Reilly SJ, Glanville EJ, Dhorepatil B, Prentice LR, Mol BW, Johnson NP. The IVF-LUBE trial - a randomized trial to assess Lipiodol(R) uterine bathing effect in women with endometriosis or repeat implantation failure undergoing IVF. Reprod Biomed Online. 2019 Mar;38(3):380-386. doi: 10.1016/j.rbmo.2018.11.015. Epub 2018 Dec 7. PMID 30679138
- [Background] Fatourechi V. Subclinical hypothyroidism: an update for primary care physicians. Mayo Clin Proc. 2009;84(1):65-71. doi: 10.4065/84.1.65. PMID 19121255